CLINICAL TRIAL: NCT06896214
Title: The Effect of Standardised Nursing Care Given to Women With Peri-Natal Loss on Peri-Natal Grief, Posttraumatic Stress, Postpartum Depression
Brief Title: The Effect of Nursing Care With Peri-Natal Loss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Canan Uçakçı Asalıoğlu, Dr., Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Canan Uçakcı Asalıoğlu; No funding support was receive (Registry Identifier: No funding support was received for this study.)
Record Dates: First submitted 2025-02-14; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Perinatal Loss; Perinatal Grief
Keywords: perinatal grief, perinatal loss,; Postpartum Depression; post-traumatic stress disorder
MeSH Terms: conditions — Depression, Postpartum; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: In this study, two of the researchers will carry out the application and the other researchers will be blinded. However, participant blinding will not be possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention(Nursing care) (Experimental): After the women are discharged, tele-nursing care will be provided by evaluating them through a telephone application that allows online interviews. In this context, three interviews will be conducted on the second day, seventh day and 15th day after discharge. EPDS will be administered on the 10th day after discharge, EPDS, I-ESR, PMS will be administered at the 1st month, 3rd month, 6th month, and prolonged grief scale (PBS) will be administered only at the 6th month. The scales will be converted into an online questionnaire and sent to the participants and will be filled in.
  Interventions: Other: Standardised nursing care intervention
- Control (Standard care) (No Intervention): Women in the control group will receive the standard care provided in the hospital. EPDS will be administered on the 10th day after discharge, EPDS, I-ESR, PMS at the 1st month, 3rd month, 6th month and prolonged grief scale (PBS) only at the 6th month. The scales will be converted into an online questionnaire and sent to the participants and will be filled in.

INTERVENTIONS:
Other: Standardised nursing care intervention — Standardised nursing care intervention
  Arms: İntervention(Nursing care)

SUMMARY:
This study was planned to evaluate the effect of standardised nursing care given to women with perinatal loss using the nursing process on perinatal grief, posttraumatic stress and postpartum depression.

H01: There is no difference between pre-test, post-test and follow-up tests in terms of perinatal grief scale mean scores in the intervention group.

H02: There is no difference between pre-test, post-test and follow-up tests in terms of IES-R mean scores in the intervention group.

H03: There is no difference between pre-test, post-test and follow-up tests in terms of EPDS mean scores in the intervention group.

H04: There is no difference between the pre-test post-test and follow-up tests in terms of the mean scores of the Complicated Grief Scale in the intervention group.

* At the first encounter with women, the mean scores of PMI, IESR and EPDS will be evaluated.
* The mean EPDS score will be evaluated on the 10th postpartum day, 1st, 3rd and 6th month.
* The mean I-ESR scale score will be evaluated at postpartum 1st, 3rd and 6th month.
* At postpartum 1st and 3rd month, the mean score of PMS will be evaluated.
* At the postpartum 6th month, the mean score of the PBI scale will be evaluated.

ELIGIBILITY:
Inclusion Criteria:- To be over 18 years old

* Being married (according to the woman's declaration)
* Not having an existing psychiatric illness (according to the woman's declaration)
* Not having communication problems (knowing Turkish, being literate, not having vision, speech or hearing problems, etc.)
* Spontaneous conception
* Singleton pregnancy
* No substance addiction

Exclusion Criteria:Women who agreed to participate in the study but did not want to receive post-discharge care, who were hospitalised for any reason, who became pregnant again, who did not want to complete the last tests or who wanted to leave the study at any stage of the study will be excluded from the sample.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women will be included in the study.
Enrollment: 58 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Peritanal grief scale | at the 1st and 3rd postpartum months. The perinatal grief scale is scored between 32-160
  - The mean PGS score will be evaluated at the 1st and 3rd postpartum months.
Edinburgh Postpartum depression scale | Postpartum day 10, 1, 3 and 6 month. The Edinburgh Postpartum Depression Scale is scored between 0 and 30.
  - The mean EPDS score will be evaluated at postpartum day 10, 1, 3 and 6 months.
Impact of Events Scale-revised | Postpartum 1, 3 and 6 months. The Impact of Events Scale is scored between 0 and 88.
  - The mean IESR score will be evaluated at 1, 3 and 6 months.
Complicated grief scale | At the 6th postpartum month.The Complicated Grief Scale is scored between 0 and 55. As the score increases, the severity of grief increases.
  At the 6th postpartum month, the mean score of the CGS will be evaluated.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol